CLINICAL TRIAL: NCT06656325
Title: An Evaluation of the Effect of the Erchonia Corporation FX-405 Laser as an Adjunctive Treatment of Periodontitis
Brief Title: An Evaluation of the Effect of the Erchonia FX-405 Laser as an Adjunctive Treatment of Periodontitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-GUM
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Periodontal Diseases; Periodontitis; Gum Disease
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Gingival Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Erchonia® FX405 (Active Comparator): The Erchonia® FX405 is made up of (3) 6405 nanometers red laser diodes and (1) 405 nanometers violet laser diode mounted in a robotic scanner device.
  Interventions: Device: Erchonia® FX405
- Placebo Laser (Placebo Comparator): The Placebo Laser has the same appearance as the Erchonia® FX405 but does not emit any therapeutic light.
  Interventions: Device: Placebo Laser

INTERVENTIONS:
Device: Erchonia® FX405 — Procedure administrations with the Erchonia® FX-405 will be applied eight times during the 5-month procedure administration phase. Phase One involves one procedure administration each week for 4 consecutive weeks. Phase 2 commences for one month following the completion of Phase One and involves one procedure administration each month for the next four consecutive months. Each procedure administration with the Erchonia FX405 takes 10 minutes and will be administered by the test site.
  Additionally, subjects will receive Scaling and Root Planing prior to the administration of the first procedure with the Erchonia FX405, and a second time at the 3-month study midpoint assessment visit.
  Arms: Erchonia® FX405
Device: Placebo Laser — Procedure administration with the Placebo Laser (emitting non therapeutic light) will be applied eight times during the 5-month procedure administration phase. Phase One involves one procedure administration each week for 4 consecutive weeks. Phase 2 commences for one month following the completion of Phase One and involves one procedure administration each month for the next four consecutive months. Each procedure administration with the Placebo Laser takes 10 minutes and will be administered by the test site.
  Additionally, subjects will receive Scaling and Root Planing prior to the administration of the first procedure with the Placebo Laser, and a second time at the 3-month study midpoint assessment visit.
  Arms: Placebo Laser

SUMMARY:
The purpose of this clinical study is to determine the effectiveness of the Erchonia® FX-405 (manufactured by Erchonia Corporation (the Company) in providing a noninvasive adjunctive treatment in combination with periodontal scaling and root planing for improving the treatment of periodontal disease.

DETAILED DESCRIPTION:
The purpose of this clinical study is to determine the effectiveness of the Erchonia® FX-405 (manufactured by Erchonia Corporation (the Company) in providing a noninvasive adjunctive treatment in combination with periodontal scaling and root planing for improving the treatment of periodontal disease. This clinical study is a double-blind design, such that neither the subject, nor the investigators - the investigator administering the treatment with the Erchonia® FX-405™ device (administration investigator) or the investigator recording the outcome measures (assessment investigator) - will be aware of whether the subject has been assigned to the active treatment test group or to the sham treatment control group until after the study is complete. All study subjects, regardless of treatment group assignment will receive active scaling and root planing standard of care therapy in addition to the active or sham therapy with the Erchonia® FX-405™ device.

ELIGIBILITY:
Inclusion Criteria:

* Subject has voluntarily signed a written informed consent form.
* Male or female 22 to 75 years of age, inclusive.
* Subject has no evidence of Localized Aggressive Periodontitis.
* Tooth loss due to periodontitis of ≤ 4 teeth.
* Two or more teeth with the following characteristics: Non 3rd molar, Periodontitis: Stage III (Severity) according to the Interdental CAL (at site of greatest loss) and RBL, as classified by the American Academy of Periodontology (AAP), No evidence of caries, No abscess infection, No previous periodontal surgery within the prior 12 months
* Subject agrees to adhere to study provided home care instructions to maintain adequate oral hygiene during the study duration.
* Subject agrees to refrain from the use of smokeless chewing tobacco for the study duration.
* Subject agrees to refrain from exceeding 40 milligrams per day of inhaled nicotine, encompassing cigarettes, electronic cigarettes, and cigars.
* Subject agrees to refrain from engaging in any other treatments for his or her periodontitis that is outside the scope of this study during his or her participation in this study

Exclusion Criteria:

* Gingival recession which may be genetic, induced secondary to orthodontic treatment, induced secondary to frenulum attachments, or present as a result of dental malocclusion.
* History of oral cancer or HIV in the last 6 months
* Pregnant or intending to become pregnant in the next 8 months.
* Sensitivity to, or contraindication for, light therapy.
* Currently enrolled in a clinical study of an investigational drug or device.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a change in Clinical Attachment Loss of ≥-2mm at the primary tooth assessment site | Baseline and 8 months
  The Clinical Attachment Loss (CAL) from baseline to endpoint (8 months) measurement is calculated for each subject. Individual subject success is defined as a 2mm or greater change in CAL at the primary tooth assessment site across the evaluation period. A negative (-) change indicates a reduction in periodontitis and is positive for individual subject success. A lower CAL score from baseline to study endpoint represents a better outcome, whereas a higher score from baseline to study endpoint represents a worse outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - 805 Dentistry, Thousand Oaks, California
  - Acton Dental Associates, Acton, Massachusetts